CLINICAL TRIAL: NCT04485481
Title: A Double-Blind, Phase 1, Single and Multiple Ascending Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of ADX-914 in Healthy Volunteers
Brief Title: Single and Multiple Ascending Dose Study of ADX-914 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Q32 Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ADX-914-001
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Safety Issues

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Cohort 1:1 - 1:6 ADX-914 (Experimental): ADX-914 single SC dose
  Interventions: Drug: ADX-914
- Placebo Comparator: Cohort 1:1 - 1:6 placebo (Placebo Comparator): Placebo single SC dose
  Interventions: Drug: Placebo
- Experimental: Cohort 2:1- 2:3 (Experimental): ADX-914 multiple SC dose once every 2 weeks for 6 weeks
  Interventions: Drug: ADX-914
- Placebo Comparator: Cohort 2:1- 2:3 (Placebo Comparator): Placebo multiple SC dose once every 2 weeks for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADX-914 — Single dose from 0.1mg/kg to TBD
  Arms: Experimental: Cohort 1:1 - 1:6 ADX-914
Drug: Placebo — Matching single dose placebo
  Arms: Placebo Comparator: Cohort 1:1 - 1:6 placebo
Drug: ADX-914 — Multiple dose from TBD to TBD
  Arms: Experimental: Cohort 2:1- 2:3
Drug: Placebo — Matching multiple dose placebo
  Arms: Placebo Comparator: Cohort 2:1- 2:3

SUMMARY:
A two (2) part study to evaluate the safety, tolerability and PK of ADX-914

DETAILED DESCRIPTION:
Part 1 - SAD:

It is expected that there will be up to 6 cohorts of 8 participants per cohort. In each cohort, participants will be randomly assigned in a 3:1 ratio to receive either ADX-914 or matching placebo.

It is planned that for each cohort in Part 1 a staggered 'sentinel' dose design will be used.

Part 2 - MAD It is expected that there will be up to 3 cohorts of 8 participants per cohort. In each cohort, participants will be randomly assigned in a 3:1 ratio to receive either ADX-914 or matching placebo. Doses will occur every 2 weeks, for a total of 4 doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the Investigator, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG recording
* Men and women age 18-50

Exclusion Criteria:

* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin levels greater than 1.5 x the upper limit of normal (ULN) at Screening or Day -1.
* QT-interval measurements corrected according to the Fridericia rule (QTcF >450 msec) during controlled rest at Screening or family history of long QT syndrome.
* Any clinically significant abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, in the judgment of the Investigator, may interfere with the interpretation of QTc-interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy.
* A clinically significant vital signs abnormality, as judged by the Investigator, at Screening, or Day -1. This includes, but is not limited to, the following, in the supine position: (a) systolic blood pressure <90 or >140 mmHg, (b) diastolic blood pressure <40 or >90 mmHg, or (c) heart rate <40 or >100 beats per minute.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Screening to end of study, up to 18 weeks
  Listing and summary of AE incidence
Number of subjects with Physical exam findings | Screening to end of study, up to 18 weeks
  Listing of clinically significant changes in PE findings
Number of subjects with Clinical safety lab changes | Screening to end of study, up to 18 weeks
  Listing and change from baseline to end of study
Number of subjects with Systolic blood pressure changes | Screening to end of study, up to 18 weeks
  Listing and change from baseline to end of study
Number of subjects with Heart rate changes | Screening to end of study, up to 18 weeks
  Listing and change from baseline to end of study
Number of subjects with 12 Lead ECG changes | Screening to end of study, up to 18 weeks
  Change in 12-lead ECG parameters from baseline to end of study

SECONDARY OUTCOMES:
Maximum observed plasma concentration, Cmax | Predose to Day 91 (SAD) and Day 127 (MAD)
  Of ADX-914
Time to reach maximum observed plasma concentration, Tmax | Predose to Day 91 (SAD) and Day 127 (MAD)
  Of ADX-914
Area Under the plasma concentration time curve, AUC | Predose to Day 91 (SAD) and Day 127 (MAD)
  Of ADX-914

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No